CLINICAL TRIAL: NCT00666068
Title: Effects of CRH on the Sleep in Patients With Hypopituitarism
Brief Title: Effects of Corticotropin Releasing Hormone (CRH) on the Sleep in Patients With Hypopituitarism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Prof. Dr. Axel Steiger, Max-Planck-Institute of Psychiatry
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: L2/2003A
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Hypopituitarism
Keywords: Patients with hypopituitarism
MeSH Terms: conditions — Hypopituitarism | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with hypopituitarism
  Cross over design: see interventions 1-2
  Interventions: Other: corticotropin releasing hormone (CRH); Other: Placebo
- 2 (Placebo Comparator): Parallel design:
  Healthy controls to be compared with placebo condition in patients with hypopituitarism
  Interventions: Other: Placebo

INTERVENTIONS:
Other: corticotropin releasing hormone (CRH) — 50 µg injected at 2200, 2300, 0000, and 0100
  Arms: 1
Other: Placebo — injected at 2200, 2300, 0000, and 0100
  Arms: 1
Other: Placebo — injected at 2200, 2300, 0000, and 0100
  Arms: 2

SUMMARY:
In contrast to healthy subjects, patients with hypopituitarism do not exhibit endocrine responses when hormones are injected. This is at least true for those with a complete insufficiency of the anterior pituitary. For example, administration of corticotropin releasing hormone (CRH) is not followed by an increase of ACTH and cortisol. Therefore, "pure" hormone effects can be investigated.

It is well established that hormones of the hypothalamic-pituitary-adrenal axis are involved in sleep regulation. In rodents, CRH decreased slow wave sleep (SWS). In humans, CRH was reported to increase wakefulness and to decrease SWS and REM sleep. Primary objective was therefore to study the effect of CRH on patients with hypopituitarism.

To date, there is no information on sleep of patients with hypopituitarism. Secondary objective is therefore to compare sleep of patients with hypopituitarism with sleep of age-matched healthy controls.

ELIGIBILITY:
Patients with hypopituitarism

Inclusion Criteria:

* Age 18-75 years
* Complete insufficiency of the anterior pituitary
* Stable hormone substitution for at least 3 months

Exclusion Criteria:

* Hormone excess in the past
* Sleep disorder, e.g. sleep apnea syndrome

Healthy controls

Inclusion Criteria:

* Age 18-75 years

Exclusion Criteria:

* Any medication during 6 week prior to study entry
* Shift work

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sleep-EEG variables, conventionally and quantitatively analyzed | within the first month

CONTACTS AND LOCATIONS:
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Germany